CLINICAL TRIAL: NCT07313371
Title: Efficacy of Clonidine in Reducing Craving in Inpatients With Cocaine/Crack Use Disorder: A Randomized Clinical Trial.
Brief Title: Efficacy of Clonidine in Reducing Craving in Inpatients With Cocaine/Crack Use Disorder
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Dângela Layne Silva Lassi, Coordinator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 86251324.2.0000.0068
Record Dates: First submitted 2025-12-02; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cocaine Use Disorder; Crack Abuse or Dependence
Keywords: crack; cocaine; craving
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Clonazepam 0,25 mg
  Interventions: Drug: clonazepam 0,25 mg
- Intervention (Experimental): Clonidine 0,1 mg
  Interventions: Drug: clonidine

INTERVENTIONS:
Drug: clonidine — Clonidine 0,1 mg bid
  Arms: Intervention
Drug: clonazepam 0,25 mg — clonazepam 0,25 mg bid
  Arms: Control

SUMMARY:
This is a single-center, randomized intervention study in a volunteer population of patients with cocaine/crack use disorder to evaluate the pharmacological treatment of cocaine/crack craving, comparing the drug clonidine with the active placebo clonazepam.

DETAILED DESCRIPTION:
Patients included will be administered clonidine 0.1 mg every 12 hours or clonazepam 0.25 mg every 12 hours for the first 2 weeks of treatment, followed by a washout for the final 2 weeks. The medication will be administered under the supervision of a member of the nursing staff. Patients will be monitored with vital signs three times a day to track changes that may be caused by the medication, such as reduced heart rate and hypotension. The primary outcome measure will be the change in cocaine craving at admission and two weeks after the start of treatment, using the visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the adult Alcohol and Drugs ward of the Perdizes Institute (IPer) at the Hospital das Clínicas, University of São Paulo Medical School
* DSM-5 criteria for cocaine and/or crack use disorder
* Voluntarily seeking treatment
* Must be able to swallow pills

Exclusion Criteria:

* Inability to read and/or understand the study questionnaires
* benzodiazepine use disorder
* opioid use disorder
* alcohol use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Daily from enrollment to end of treatment at 2 weeks; then after 30, 60 and 90 days after end of treatment
  Visual Analog Scale for craving, ranging from 0 to 10, where 0 means no craving and 10 means maximum craving

SECONDARY OUTCOMES:
Adverse Effects | from the beginning of the intervention to 90 days after enrollment in the study
  Spontaneous reports
Blood pressure | Three times daily from baseline up to 14 days
  Diastolic and systolic pressure in mmHg
Heart Rate | Three times daily from baseline up to 14 days
  Heart rate in beats per minute
Cinical Global Impression - Severity of Illness (CGI-S) | At baseline
  The Clinical Global Impression - Severity of Illness (CGI-S) is a brief, clinician-rated scale used to assess the current severity of a patient's mental illness at the time of assessment, ranging from 1 (1 Normal, not at all ill) to 7 (Among the most extremely ill patients)
Clinical Global Impression - Improvement (CGI-I) | Will be assessed after 1 and 2 weeks from baseline
  The Clinical Global Impression - Improvement (CGI-I) scale is a single-item, clinician-rated assessment tool used to measure the change in a patient's overall clinical condition since the baseline, ranging from 1 (very much improved) to 7 (Very much worse)
Crack/Cocaine Use | 30, 60 and 90 days after the end of the intervention
  The Timeline Followback (TFLB) will be used to measure the patient's average daily drug use in standardized units (e.g. Units, grams, or rocks of cocaine/crack)

CONTACTS AND LOCATIONS:
Overall Officials: Dangela L S Lassi, Principal Investigator — Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roque Bravo R, Faria AC, Brito-da-Costa AM, Carmo H, Mladenka P, Dias da Silva D, Remiao F, On Behalf Of The Oemonom Researchers. Cocaine: An Updated Overview on Chemistry, Detection, Biokinetics, and Pharmacotoxicological Aspects including Abuse Pattern. Toxins (Basel). 2022 Apr 13;14(4):278. doi: 10.3390/toxins14040278. PMID 35448887
- See also: United Nations Office on Drugs and Crime. Treatment of Stimulant Use Disorders: Current Practices and Promising Perspectives. — https://www.unodc.org/unodc/data-and-analysis/world-drug-report-2022.html
- See also: Drug Misuse and Addiction. National Institute on Drug Abuse website — https://nida.nih.gov/publications/drugs-brains-behavior-science-addiction/drug-misuse-addiction